CLINICAL TRIAL: NCT00564213
Title: Evaluation of the Prophylactic Use of Mitomycin C 0.02% to Inhibit Haze Formation After Photorefractive Keratectomy for High Myopia: 15 x 30 Seconds
Acronym: BQ-01-07-ARVO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Olhos de Goiania (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BQ -1-07-ARVO
Record Dates: First submitted 2007-11-26; First posted 2007-11-27 (Estimated); Last update posted 2008-11-26 (Estimated); Status verified 2007-11

CONDITIONS: High Myopia
Keywords: Myopia; Mitomycin
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): A single intraoperative topical application of mitomycin C 0.02% for 15 seconds
  Interventions: Drug: PRK and a single intraoperative topical application of mitomycin C 0.02% for 15 seconds
- 2 (Experimental): A single intraoperative topical application of mitomycin C 0.02% for 30 seconds
  Interventions: Drug: PRK and a single intraoperative topical application of mitomycin C 0.02% for 15 seconds

INTERVENTIONS:
Drug: PRK and a single intraoperative topical application of mitomycin C 0.02% for 15 seconds — Mitomycin 0.02%

SUMMARY:
To evaluate and compare the effect of the prophylactic use of two different exposure times of mitomycin C (MMC) 0.02% to inhibit haze formation after photorefractive keratectomy (PRK) for high myopia (> -7.0 D).

Methods: Forty six eyes of twenty three patients, 8 men and 15 women, with high myopia were included in this prospective study. Mean age at the time of PRK plus MMC was 31.7 years. Before PRK, the mean spherical equivalent was -8.50 D (range, -7.25 to -10.50 D). In each patient, one eye was randomly assigned to PRK and a single intraoperative topical application of mitomycin C 0.02% for 15 seconds (Group 1) and the fellow eye, for 30 seconds (Group 2).The inclusion criteria were high myopia, no central corneal opacity and inadequate corneal thickness to allow a safe Laser in situ keratomileusis procedure. Refraction, uncorrected visual acuity, best spectacle-corrected visual acuity (BSCVA), and slit-lamp evidence of corneal opacity (haze) were evaluated over 12 months

ELIGIBILITY:
Inclusion Criteria:

* Myopia or compound myopic astigmatism
* Stable refractive error
* No associated eye disease

Exclusion Criteria:

* Diabetes,
* Autoimmune diseases
* Topographic abnormalities

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2005-03; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Belquiz A Nassaralla, Study Chair — Instituto de Olhos de GOiânia